CLINICAL TRIAL: NCT01966276
Title: Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Methylphenidate Hydrochloride as a Treatment for Chronic Fatigue Syndrome in Patients Taking a CFS-Specific Nutrient Formula
Brief Title: The Synergy Trial: Methylphenidate Plus a CFS-Specific Nutrient Formula as a Treatment for Chronic Fatigue Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: K-PAX Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KPAX-002-01
Record Dates: First submitted 2013-10-14; First posted 2013-10-21 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Fatigue Syndrome (CFS); Myalgic Encephalomyelitis (ME)
Keywords: Chronic Fatigue Syndrome (CFS); Myalgic Encephalomyelitis (ME); central nervous system (CNS); fatigue; alertness; brain fog; mitochondria; methylphenidate; Ritalin; stimulant; multivitamin; multimineral; micronutrients; supplements
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Mental Fatigue | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methyl-P plus Nutrient Formula (Experimental): Methylphenidate hydrochloride plus a CFS Nutrient Formula, both taken twice daily.
  The CFS Nutrient Formula is a broad-spectrum CFS-specific dietary supplement that provides CFS patients with cellular fuel and cofactors (amino acids, antioxidants, and mitochondrial cofactors) while the low-dose CNS stimulant (methylphenidate hydrochloride) provides a metabolic catalyst to enhance cellular metabolism.
  Interventions: Drug: Methyl-P plus Nutrient Formula
- Methyl-P plus Nutrient matched placebos (Placebo Comparator): Methylphenidate matched placebo + CFS Nutrient Formula matched placebo, both taken twice daily.
  Interventions: Drug: Methyl-P plus Nutrient matched placebos

INTERVENTIONS:
Drug: Methyl-P plus Nutrient Formula — * Week 1 (take the following together twice a day-at breakfast and lunch)
    * One tablet of Methyl-P (5mg)
    * Four tablets of CFS Nutrient Formula
  * Week 2 to Week 12 (take the following together twice a day-at breakfast and lunch):
    * Two tablets of Methyl-P (10mg)
    * Four tablets of CFS Nutrient Formula
  Other Names: Ritalin
  Arms: Methyl-P plus Nutrient Formula
Drug: Methyl-P plus Nutrient matched placebos — * Week 1 (take the following together twice a day-at breakfast and lunch)
    * One tablet of Methyl-P Placebo
    * Four tablets of CFS Nutrient Placebo
  * Week 2 to Week 12 (take the following together twice a day-at breakfast and lunch):
    * Two tablets of Methyl-P Placebo
    * Four tablets of CFS Nutrient Placebo
  Arms: Methyl-P plus Nutrient matched placebos

SUMMARY:
The Synergy Trial will evaluate the safety and efficacy of a currently available medication (methylphenidate hydrochloride) combined with a CFS-specific dietary supplement (CFS Nutrient Formula) to treat Chronic Fatigue Syndrome (CFS).

DETAILED DESCRIPTION:
The Synergy Trial will evaluate the safety and efficacy of a currently available medication (methylphenidate) combined with a CFS-specific dietary supplement (CFS Nutrient Formula) to treat Chronic Fatigue Syndrome (CFS).

The CFS Nutrient Formula to be used in this trial is a broad-spectrum micronutrient supplement that provides CFS patients with vitamins, minerals, and other cofactors (amino acids, antioxidants, and mitochondrial cofactors) to complement the low-dose Central Nervous System (CNS) stimulant (methylphenidate). In other words, therapeutic dosages of micronutrients are provided to support the functioning of the nervous, endocrine, and immune systems to a level at which a lower than customary dosage of methylphenidate can produce positive clinical effects on CFS symptoms and also be well tolerated.

Methylphenidate is the generic form of Ritalin®. The dose being tested in this study is relatively low (5-10mg twice daily). This drug has been in clinical use for over 50 years for the treatment of Narcolepsy and Attention Deficit Disorder and has a well-described safety profile when used as recommended. Methylphenidate alone has been studied as a treatment for CFS in the past and has been shown to produce mild benefits and be well-tolerated. When provided as innovative therapy, methylphenidate plus this CFS Nutrient Formula has produced substantial improvements in CFS symptoms in a limited number of patients, and demonstrated excellent tolerability.

Use of low dose methylphenidate hydrochloride coadministered with a CFS Nutrient Formula has not been previously evaluated in a controlled clinical study. The risk to patients using this combination is believed to be low, especially in the context of a well-controlled clinical study. Furthermore, this combination is not expected to increase the incidence or severity of adverse events associated with methylphenidate hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must fulfill the 1994 CDC case definition of CFS (Fukuda et al., Ann Intern Med. 1994; 121:953-959)
* Subjects must also report alertness and/or concentration deficits
* Otherwise in good health based on medical history and screening evaluation
* Willingness to NOT take any nutritional or herbal supplements other than the study treatment during the course of the trial
* Nutritional supplements that are exempted from this requirement are limited to the following:

  * Probiotic supplements
  * Fiber supplements
  * Fish oil supplements
  * Digestive enzymes
  * Melatonin ≤ 10mg per day
  * Calcium ≤ 600 mg per day
  * Magnesium ≤ 400 mg per day
  * Vitamin D ≤ 400 i.u. per day
* Willingness to NOT consume any caffeine-containing supplements during the study period (coffee, tea, or chocolate are exempt). These include but are not limited to the following beverages:

  * Red Bull®
  * Monster®
  * Rockstar®
  * 5-hour® energy shots
* Willingness to NOT consume any pseudoephedrine-containing products during the study period
* Willingness to practice effective contraception

Exclusion Criteria:

* Pregnancy or lactation
* Active substance abuse
* Major depression as defined by Zung Depression Scale score ≥ 60
* Use of rintatolimod (Ampligen®) within the past 3 months
* Currently taking any prescription medication to treat anxiety on a daily basis
* Use of more than 3 times/week within the past 3 months of:

  * Monoamine oxidase inhibitors (MAOs)
  * Anti-psychotic medications
  * CNS stimulants (i.e. Provigil®, Nuvigil®, Adderall®, Ritalin®, amphetamines)
  * Narcotic opioids
  * Tramadol (i.e. Ultram®, Ultracet®, Conzip®, or Ryzolt®)
  * Gabapentin (Neurontin®) > 600mg/day
  * Pregabalin (Lyrica®)
  * Duloxetine (Cymbalta®)
  * Milnacipran (Savella®)
  * Coumarin anticoagulants (Coumadin®)
  * Valganciclovir (Valcyte®)
* Daily concurrent use of more than one antidepressant medication except if one of the two antidepressant medications are:

  * Amitriptyline ≤ 30mg at bedtime
  * Trazodone ≤ 50mg at bedtime
  * Doxepin ≤ 20mg at bedtime
* Active medical conditions to which treatment with methylphenidate hydrochloride or micronutrients may be contraindicated, including:

  * Glaucoma
  * Diabetes Mellitus
  * Current stomach or duodenal ulcer
  * Uncontrolled hypertension (blood pressure at screening of systolic >150 or diastolic >90)
  * Heart disease (including cardiac arrhythmia, cardiac ischemia, syndrome of Gilles de la Tourette or a past history of myocardial infarction or cerebrovascular event)
  * Motor tics or family history of psychosis or bipolar disorder
  * Previous history or seizures
* A diagnosis of other conditions that may be in part responsible for the patient's fatigue including, but not limited to:

  * HIV infection
  * Chronic Hepatitis B & C
  * Cancer (receiving treatment either currently or within the past two years)
  * Chronic Renal Disease
* Clinically significant laboratory test values as determined by the Investigator
* Clinically significant ECG abnormalities as determined by the Medical Monitor
* Compliance criteria: A subject will not be eligible if he/she, in the opinion of the Investigator, will be unable to comply with any aspect of this study protocol, including the visit schedule.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported Checklist Individual Strength (CIS) Total Score | Week 12

SECONDARY OUTCOMES:
Percentage of patients with 20% or greater improvement in the CIS total score | Week 12
Concentration Disturbances Subscore on the CIS | Week 12
Concentration Disturbances Score by Visual Analog Scale (VAS) | Week 12
Fatigue Score by Visual Analog Scale (VAS) | Week 12
Pain Symptoms by Brief Pain Inventory Form | Week 12
Patient Global Assessment of Change Questionnaires (for Fatigue and Sleep) | Week 12
Number of Participants with Adverse Events to Assess Safety and Tolerability | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jose Montoya, M.D., Principal Investigator — Stanford University School of Medicine, Division of Infectious Diseases
Locations (4):
- United States (4):
  - Stanford Chronic Fatigue Syndrome/ME Initiative, Stanford, California
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Susan Levine, MD, New York, New York
  - Fatigue Consultation Clinic, Salt Lake City, Utah